CLINICAL TRIAL: NCT06287944
Title: Phase I Study of Escalating Doses of 225Ac-DOTA-Anti-CD38 Daratumumab Monoclonal Antibody Added to the Conditioning Regimen of Fludarabine, Melphalan and Organ Sparing Total Marrow and Lymphoid Irradiation (TMLI) as Conditioning for Allogeneic Hematopoietic Cell Transplantation in Patients With High-Risk Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia and Myelodysplastic Syndrome
Brief Title: 225Ac-DOTA-Anti-CD38 Daratumumab Monoclonal Antibody With Fludarabine, Melphalan and Total Marrow and Lymphoid Irradiation as Conditioning Treatment for Donor Stem Cell Transplant in Patients With High-Risk Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia and Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23694; NCI-2024-01131 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23694 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-02-16; First posted 2024-03-01 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Specimen Handling; Biopsy; daratumumab; fludarabine; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Indium; Melphalan; Nuclear Medicine Department, Hospital; X-Rays; Photons; Sirolimus; Tacrolimus; Lymphatic Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment ( Actinium Ac 225-DOTA-Daratumumab) (Experimental): Patients receive daratumumab IV over 45 minutes followed by indium In 111-DOTA-daratumumab IV over 15 minutes and actinium Ac 225-DOTA-daratumumab IV over ~20-40 minutes on day -15. Patients receive TMLI BID on days -8 to -5, fludarabine IV on days -4 to -2 and melphalan IV on day -2, followed by HCT on day 0. Patients receive GVHD prophylaxis with sirolimus and tacrolimus starting on day -1. Patients also undergo CT during screening, nuclear scan and SPECT scans on study, bone marrow biopsy and aspiration, echocardiography, or MUGA, and blood sample collection during screening and throughout study.
  Interventions: Biological: Actinium Ac 225-DOTA-Daratumumab; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Biological: Daratumumab; Procedure: Echocardiography; Drug: Fludarabine; Procedure: Hematopoietic Cell Transplantation; Biological: Indium In 111-DOTA-Daratumumab; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Procedure: Radionuclide Imaging; Procedure: Single Photon Emission Computed Tomography; Drug: Sirolimus; Drug: Tacrolimus; Radiation: Total Marrow and Lymphoid Irradiation

INTERVENTIONS:
Biological: Actinium Ac 225-DOTA-Daratumumab — Given IV
  Other Names: 225Ac-DOTA-Daratumumab; [225Ac]-DOTA-Daratumumab
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Biological: Daratumumab — Given IV
  Other Names: Daratumumab Biosimilar HLX15; Daratumumab-fihj; Darzalex; HLX15; HuMax-CD38; JNJ-54767414
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Hematopoietic Cell Transplantation — Undergo SCT
  Other Names: HCT; Hematopoietic Stem Cell Infusion; Hematopoietic Stem Cell Transplantation; HSCT; SCT; Stem Cell Transplant; stem cell transplantation; Stem Cell Transplantation, NOS
Biological: Indium In 111-DOTA-Daratumumab — Given IV
  Other Names: 111In-DOTA-Daratumumab; [111In]-DOTA-Daratumumab
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Radionuclide Imaging — Undergo nuclear scan
  Other Names: NM; Nuclear Medicine; nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; Scintigraphy
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT scan
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Drug: Sirolimus — Given sirolimus
  Other Names: AY 22989; RAPA; Rapamune; Rapamycin; SILA 9268A; WY-090217
Drug: Tacrolimus — Given tacrolimus
  Other Names: FK 506; FK-506; Fujimycin; Hecoria; Prograf; Protopic; Tacforius
Radiation: Total Marrow and Lymphoid Irradiation — Undergo TMLI
  Other Names: TMLI

SUMMARY:
This phase I trial tests the safety, side effects, best dose, and effectiveness of 225Ac-DOTA-Anti-CD38 daratumumab monoclonal antibody in combination with fludarabine, melphalan and total marrow and lymphoid irradiation (TMLI) as conditioning treatment for donor stem cell transplant in patients with high-risk acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL) and myelodysplastic syndrome (MDS). Daratumumab is in a class of medications called monoclonal antibodies. It binds to a protein called CD38, which is found on some types of immune cells and cancer cells. Daratumumab may block CD38 and help the immune system kill cancer cells. Radioimmunotherapy is treatment with a radioactive substance that is linked to a monoclonal antibody, such as daratumumab, that will find and attach to cancer cells. Radiation given off by the radioisotope my help kill the cancer cells. Chemotherapy drugs, such as fludarabine and melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. TMLI is a targeted form of body radiation that targets marrow, lymph node chains, and the spleen. It is designed to reduce radiation-associated side effects and maximize therapy effect. Actinium Ac 225-DOTA-daratumumab combined with fludarabine, melphalan and TMLI may be safe, tolerable, and/or effective as conditioning treatment for donor stem cell transplant in patients with high-risk AML, ALL, and MDS.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Describe toxicities attributable to actinium Ac 225-DOTA-daratumumab (225Ac-DOTA-anti-CD38 daratumumab) radioimmunotherapy by dose level in patients treated under this regimen.

II. Determine the maximum tolerated dose/recommended phase II dose (MTD/RP2D) of 225Ac-DOTA-anti-CD38 daratumumab radioimmunotherapy with fixed doses of organ sparing TMLI (12 Gy), fludarabine and melphalan (FM100) as conditioning regimen for allogeneic hematopoietic cell transplantation (HCT) for treatment of high-risk acute myeloid leukemias, acute lymphoblastic leukemia or myelodysplastic syndrome (MDS), in patients who are not eligible for standard myeloablative regimens.

SECONDARY OBJECTIVES:

I. Evaluate the safety of the regimen, at each dose level, by assessing the following:

Ia. Type, frequency, severity, attribution, time course and duration of adverse events, including acute/chronic graft-versus-host disease (GVHD), infection and delayed engraftment.

II. Estimate overall survival (OS), event-free survival (EFS), GVHD relapse free survival (GRFS), cumulative incidence (CI) of relapse/progression, and non-relapse mortality (NRM) at 100 days, 1 year and 2 years.

III. Describe biodistribution, pharmacokinetics and organ dosimetry of 225Ac-DOTA-daratumumab.

OUTLINE: This is a dose escalation of actinium Ac 225-DOTA-Daratumumab in combination with fludarabine, melphalan and TMLI.

Patients receive daratumumab intravenously (IV) over 45 minutes followed by indium In 111-DOTA-daratumumab IV over 15 minutes and actinium Ac 225-DOTA-daratumumab IV over ~20-40 minutes on day -15. Patients receive TMLI twice daily (BID) on days -8 to -5, fludarabine IV on days -4 to -2 and melphalan IV on day -2, followed by HCT on day 0. Patients receive GVHD prophylaxis with sirolimus and tacrolimus starting on day -1. Patients also undergo computed tomography (CT) during screening, nuclear scan and single photon emission computed tomography (SPECT) scans on study, bone marrow biopsy and aspiration, echocardiography, or multigated acquisition scan (MUGA), and blood sample collection during screening and throughout study.

After completion of study treatment, patients are followed up twice weekly for the first 100 days post-transplant, then twice monthly up to 6 months post-transplant followed by monthly until discontinuation of immunosuppressive therapy without evidence of GVHD with at least yearly follow-up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* ≥ 60 years. Note: Patients ≥ 18 years and < 60 years with HCT-comorbidity index (CI) ≥ 2 are also included
* Karnofsky performance status ≥ 70
* Eligible patients will have a histopathological confirmed diagnosis of hematologic malignancy in one of the following categories :

  * Acute myelogenous leukemia:

    * Patients with de novo or secondary disease in unfavorable risk group including poor risk cytogenetics according to National Comprehensive Cancer Network (NCCN) guidelines for AML i.e., monosomal karyotype, -5,5q-,-7,7q-,11q23-non t(9;11), inv (3), t(3;3), t(6;9), t(9;22) and complex karyotypes (≥ 3 unrelated abnormalities), or all patient in intermediate risk groups accept patients with FLT3-NPM1+ disease, OR
    * Patients with a complete morphological remission (CR) with minimal residual disease (MRD)-positive status by flow cytometry (≥ 0.1% by flow cytometry) or cytogenetic after at least 2 prior induction therapies, OR
    * Patients with chemosensitive active disease defined as at least 50% reduction in their blast count after last treatment
  * Myelodysplastic syndrome in high-intermediate (int-2) and high-risk categories per Revised International Prognostic Scoring System- (IPSS-R)
  * Acute lymphocytic leukemia

    * Patients with de novo or secondary disease according to NCCN guidelines for ALL hypoploidy (< 44 chromosomes); t(v;11q23): MLL rearranged; t(9;22) (q34;q11.2); complex cytogenetics (5 or more chromosomal abnormalities); high white blood cell (WBC) at diagnosis (≥ 30,000 for B lineage or ≥ 50,000 for T lineage); iAMP21loss of 13q, and abnormal 17p, OR
    * Patients with a complete response (CR) with MRD-positive status by flow cytometry (≥ 0.1% by flow cytometry) or cytogenetics after at least 2 prior induction therapies, OR
    * Patients with chemosensitive active disease defined as at least 50% reduction in their blast count after last treatment
* A pretreatment measured creatinine clearance (absolute value) of ≥ 60 ml/minute (To be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Patients must have a serum bilirubin ≤ 2.0 mg/dl (To be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Patients must have a serum glutamic oxaloacetic transaminase (SGOT) ≤ 2.5 times the institutional upper limits of normal (To be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Patients must have a serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 times the institutional upper limits of normal (To be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Ejection fraction measured by echocardiogram or multigated acquisition scan (MUGA) ≥ 50% (To be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Diffusion capacity of the lung for carbon monoxide (DLCO) > 50% predicted (To be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Forced expiratory volume in 1 second (FEV1) > 50% predicted (To be performed within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* DONOR SPECIFIC CRITERIA: All candidates for this study must have an human leukocyte antigen (HLA) (A, B, C, and DR) identical sibling who is willing to donate mobilized peripheral blood stem cells (preferred) or bone marrow, or have a 10/10 (A, B, C, DR and DQ) allele matched unrelated donor. DQ or DP mismatch is allowed per discretion of the principal investigator. City of Hope (COH) standards of practice (SOP) (B.001.11) will be used for allogeneic donor evaluation, selection, and consent. Donor screening will be in compliance with all requirements of Food and Drug Administration (FDA) regulation 21 CFR Part 1271 including donor screening for COVID-19 exposure or infection

Exclusion Criteria:

* Patients who had a prior allogeneic transplant
* All patients with prior radiation treatment to the lung, liver, and kidney
* Patients who have received prior radiopharmaceutical therapy
* Inclusion of other patients with previous radiation exposure will be determined based on the radiation oncologist medical doctor (MD) principal investigator (PI) evaluation and judgement
* For patients with leukemia or MDS: Patients may not have received more than 3 prior regimens, where the regimen intent was to induce remission
* Receiving any other investigational agents or concurrent biological, intensive chemotherapy or radiation therapy for the previous 2 weeks from conditioning
* Patients should have discontinued all previous intensive therapy, chemotherapy, or radiotherapy for 2 weeks prior to commencing therapy on this study. Note: Low dose chemotherapy or maintenance chemotherapy given within 7 days of planned study enrollment is permitted. These include hydroxyurea, 6-meraptopurine, oral methotrexate, vincristine, oral etoposide, and tyrosine kinase inhibitors (TKIs). FLT-3 inhibitors can also be given up to 3 days before conditioning regimen
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Patients with other active malignancies are ineligible for this study, other than non-melanoma skin cancers
* Patients should not have any uncontrolled illness including ongoing or active bacterial, viral or fungal infection
* The recipient has a medical problem or neurologic/psychiatric dysfunction which would impair his/her ability to be compliant with the medical regimen and to tolerate transplantation or would prolong hematologic recovery which in the opinion of the investigator (treating physician) would place the recipient at unacceptable risk
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-05-19 (Estimated); Study Completion 2028-05-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (CTCAE) | Up to 2 years post-transplant
  Toxicity will be scored on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5 scale. Toxicity will be recorded in each patient and will include the type, severity, and probable association with the study regimen.
Incidence of adverse events (Bearman) | Up to 2 years post-transplant
  Toxicity will be scored on the Bearman Scale. Toxicity will be recorded in each patient and will include the type, severity, and probable association with the study regimen.
Dose limiting toxicity (DLT) | Up to 30 days post-stem cell infusion
  DLT will be graded using the NCI CTCAE v5 scale.
Maximum tolerated dose/recommended phase II dose (MTD/RP2D) | Up to 30 days post stem cell infusion
  MTD/RP2D will be defined as the highest dose where 6 patients have been treated and at most on patient experiences a DLT.

SECONDARY OUTCOMES:
Overall survival (OS) | At start of protocol therapy to death or last follow-up up to 2 years post transplant
  OS will be defined as the time from start of protocol therapy to death or last follow-up whichever comes first. OS will be calculated using the Kaplan-Meier method.
Event-free survival (EFS) | At start of protocol therapy to death, relapse/progression or last follow-up up to 2 years post-transplant
  EFS will be defined as the time from start of protocol therapy to death, relapse/progression or last follow-up, whichever comes first. EFS will be calculated using the Kaplan-Meier method.
Cumulative incidence of relapse/progression (CIR) | At start of therapy up to 2 years post transplant
  CIR will be measured from start of therapy. Death without relapse/progression is considered a competing risk.
Graft versus host disease and relapse free survival (GRFS) | At start of therapy up to 2 years post-transplant
  GRFS will be measured from the start of therapy. GRFS will be calculated using the Kaplan-Meier method.
Complete remission (CR) proportion | At start of therapy up to day 30
  CR will be defined as the time from start of therapy to the time of biopsy proven CR.
Non-relapse mortality (NRM) | At start of therapy until non-disease related death or last follow-up up to 2 years post-transplant
  NRM will be defined as the time from start of therapy until non-disease related death, or last follow-up, whichever comes first. NRM will be calculated as competing risks.
Incidence of infection | At day 0 up to 100 days post-transplant
  Microbiologically documented infections will be reported by site of disease, date of onset, severity and resolution, if any.
Neutrophil recovery rate | At stem cell infusion up to the first to three consecutive days with neutrophil count greater than 0.5 x 10^9/L up to 2 years post-transplant
  Neutrophil recovery rate will be measured from stem cell infusion to the first to three consecutive days with neutrophil count greater than 0.5 x 10^9/L.
Incidence of grade 2-4 and 3-4 acute graft-versus-host disease (GVHD) | At date of stem cell infusion to document/biopsy proven acute GVHS onset (within first 100 days post-transplant)
  Documented/biopsy proven acute GVHD will be graded according to the Consensus Grading. Acute GVHD will be measured from date of stem cell infusion to document/biopsy proven acute GVHD onset date (within the first 100 days post-transplant) and will be used to estimate the cumulative incidence. GVHD will be calculated as competing risks.
Incidence of chronic GVHD (cGVHD) | At 80-100 days post-transplant to documented/biopsy proven cGVHD onset date up to 2 years post-transplant
  Documented/biopsy proven cGVHD is scored according to National Institutes of Health Consensus Staging. CGVHD is measured from approximately 80-100 days post-transplant to the documented/biopsy proven cGVHD onset date and will be used to estimate the cumulative incidence. The incidence of cGVHD will be calculated as competing risks.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Y Wong, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States